CLINICAL TRIAL: NCT00760864
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of Oral TAK-715 in the Treatment of the Signs and Symptoms of Rheumatoid Arthritis
Brief Title: Safety and Efficacy of TAK-715 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-03-TL-715-005; 2004-002157-30 (EudraCT Number); U1111-1114-2984 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Drug Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(4-(2-ethyl-4-(3-methylphenyl)-1,3-thiazol-5-yl)-2-pyridyl)benzamide; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TAK-715 25 mg BID (Experimental)
  Interventions: Drug: TAK-715 and methotrexate
- TAK-715 50 mg BID (Experimental)
  Interventions: Drug: TAK-715 and methotrexate
- TAK-715 100 mg BID (Experimental)
  Interventions: Drug: TAK-715 and methotrexate
- Methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: TAK-715 and methotrexate — TAK-715 25 mg, tablets, orally, twice daily and methotrexate stable dose for up to 6 weeks.
  Arms: TAK-715 25 mg BID
Drug: TAK-715 and methotrexate — TAK-715 50 mg, tablets, orally, twice daily and methotrexate stable dose for up to 6 weeks.
  Arms: TAK-715 50 mg BID
Drug: TAK-715 and methotrexate — TAK-715 100 mg, tablets, orally, twice daily and methotrexate stable dose for up to 6 weeks.
  Arms: TAK-715 100 mg BID
Drug: Methotrexate — TAK-715 placebo-matching, tablets, orally, twice daily and methotrexate stable dose for up to 6 weeks
  Arms: Methotrexate

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TAK-715, twice daily (BID), in the treatment of rheumatoid arthritis signs and symptoms in patients with a partial response to methotrexate.

DETAILED DESCRIPTION:
Rheumatoid arthritis affects approximately 1% of the adult population, and is a chronic, progressive disease characterized by synovial inflammation. The resulting inflammation leads to destruction of the synovium and surrounding joint tissues, which can result in cartilage destruction, bone erosion and resultant loss of joint function. It is an autoimmune disorder of unknown etiology and typically affects the joints of the hand, wrist, knee, and foot, usually in a bilateral pattern. Symptoms experienced early in the disease process include pain, swelling, and tenderness of affected joints. As the disease progresses, many patients experience joint stiffness, weakness, fatigue, anorexia, and weight loss, and ultimately tissue damage and joint destruction. The severity of symptoms varies widely, ranging from annoyance to debilitation. Rheumatoid arthritis is a disease that primarily afflicts adults, with women being affected more often than men. Because rheumatoid arthritis is both chronic and destructive, it requires early diagnosis and aggressive treatment to minimize the morbidity associated with its progression, which can lead to deterioration in physical function and psychological and social well-being. The objectives of rheumatoid arthritis therapy are to reduce inflammation and to decrease the progression of articular damage. Disease-modifying antirheumatic drugs are used to accomplish these objectives.

During the past several years, rheumatologists have become increasingly aggressive in initiating treatment with disease-modifying antirheumatic drugs early in the course of rheumatoid arthritis in an attempt to prevent joint destruction. The gold standard of therapy has been methotrexate, which has been shown to be efficacious and safe, and appears to remain effective, even after many years of treatment. However, not all patients respond to methotrexate, and even patients who do respond most frequently have only a partial response (reduced signs and symptoms, but still active disease). As a result, many patients are treated with 2 or more disease-modifying antirheumatic drugs at the same time.

More recently, biologics (biotechnology drugs) have been introduced in the armamentarium against rheumatoid arthritis, based on an improved understanding of the role of the proinflammatory mediators, TNF-alpha, interleukin-1, and interleukin-6 in rheumatoid arthritis. Etanercept (Enbrel®), a soluble TNF-alpha type II receptor-human immunoglobulin fusion protein administered subcutaneously twice a week, infliximab (Remicade®), a chimeric human mouse monoclonal antibody against TNF-alpha, administered intravenously every 4 to 8 weeks along with weekly methotrexate, and adalimumab (Humira®), a human-derived recombinant immunoglobulin monoclonal antibody, administered subcutaneously every other week, are currently available for treatment of rheumatoid arthritis. They have demonstrated rapid and substantial improvement in rheumatoid arthritis, presumably by preventing the actions of TNF-alpha in the joint, thereby reducing the inflammatory and destructive consequences of TNF-alpha. Etanercept and infliximab have been granted Food and Drug Administration (FDA) approved indications for reducing signs and symptoms, inhibiting the progression of structural damage and improving physical function of patients with moderately to severely active rheumatoid arthritis. Adalimumab has been granted FDA approved indications for reducing signs and symptoms and inhibiting the progression of structural damage, and Anakinra (Kineret®), an interleukin-1 receptor antagonist administered subcutaneously daily, received FDA approval for reducing signs and symptoms.

TAK-715 is a p38 mitogen-activated protein kinase inhibitor that has shown in nonclinical studies to decrease proinflammatory cytokine production, specifically tumor necrosis factor-α (TNF-α), interleukin (IL)-1, and IL-6. These cytokines are thought to be pivotal mediators of inflammation and the resultant joint destruction in rheumatoid arthritis. TAK-715 has also been shown to inhibit the production of cyclooxygenase-2-mediated prostanoids and nitric oxide as well as oppose the differentiation of osteoclasts, each of which contributes to the joint damage associated with rheumatoid arthritis.

Individuals who participate in this study will provide written informed consent and will be required to commit to a screening visit and up to approximately 5 additional visits at the study center. Study participation is anticipated to be up to 6 months. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations and electrocardiograms. Participants will be required to provide detailed medical histories related to rheumatoid arthritis and complete multiple questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Had a diagnosis of rheumatoid arthritis using American College of Rheumatology criteria of at least 6 months duration.
* A female subject of childbearing potential who is sexually active must agree to use adequate contraception, and must be neither pregnant nor lactating from Screening throughout the duration of the study.
* Had a physical examination at Screening that revealed no clinically significant abnormalities (other than rheumatoid arthritis) in the investigator's opinion.
* Had clinical laboratory test results at Screening that were normal or, if abnormal, were not clinically significant in the investigator's opinion.
* Had a 12-lead electrocardiogram at Screening that was normal or, if abnormal, was not clinically significant in the investigator's opinion.
* Had a chest x-ray within 6 months prior to or during the Pretreatment Period that, in the investigator's opinion, showed no signs of active tuberculosis and was free of clinically significant findings.
* Had a negative purified protein derivative skin test for tuberculosis (less than or equal to 5 mm in duration) during the Screening Period.
* Had been receiving oral or parenteral methotrexate for at least 6 months prior to Baseline and must have been on a stable dose (12.5 to 25 mg per week, inclusive) of methotrexate for at least 4 weeks prior to Baseline. The subject must have been on a dose of folic acid at greater than or equal to 1 mg/day.
* Had at least 6 swollen and 9 tender joints using the 66/68 joint count scale at Screening and Baseline.
* At Screening, the subject must have had a C-reactive protein of at least 1.2 mg/dL or an erythrocyte sedimentation rate of at least 28 mm/hr.
* For individuals who were taking a systemic corticosteroid, the maintenance dose of prednisone, or its equivalent, could not exceed 10 mg/day and must have been stable for at least 4 weeks prior to Baseline and must have remained at that stable dose throughout the study.
* For individuals who were taking a nonsteroidal anti-inflammatory drug for the treatment of rheumatoid arthritis, the maintenance dose of the nonsteroidal anti-inflammatory drug must have been stable for at least 4 weeks prior to Baseline and must have remained at that stable dose throughout the study.

Exclusion Criteria:

* Had been diagnosed with any type of arthritis at age 16 or younger.
* Had a history of a clinically significant illness, medical condition, or laboratory abnormality within 3 months prior to Baseline that, in the investigator's opinion, would preclude the subject's participation in the study.
* Had a known history of human immunodeficiency virus infection.
* Had a known history of hepatitis B or C.
* Had uncontrolled hypertension.
* Had moderate or severe liver disease at Screening, as defined by at least 1 of the following conditions:

  * Aspartate transaminase or alanine transaminase greater than 1.2 times the upper limit of normal.
  * Total bilirubin greater than 1.2 times upper limit of normal (excluding subjects diagnosed with Gilbert's disease).
  * Alkaline phosphatase greater than 1.5 times upper limit of normal.
* Had elevated serum creatinine level for age and gender at Screening.
* Had hemoglobin less than 9.0 g/dL, white blood cell count of less than 3000/mm3, or a platelet count less than 100,000/mm3 at Screening.
* Had an American College of Rheumatology revised rheumatoid arthritis functional status of IV at Screening.
* Had taken, is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * A disease-modifying antirheumatic drug or a biologic agent other than methotrexate in the 8 weeks prior to Baseline, including:

    * Plaquenil.
    * Sulfasalazine.
    * Tetracycline.
    * infliximab (Remicade®).
    * leflunomide (Arava®).
    * etanercept (Enbrel®).
    * anakinra (Kineret®).
  * Had failed therapy due to lack of efficacy with any anti- tumor necrosis factor agent.
  * Had failed due to lack of efficacy with more than 2 disease-modifying antirheumatic drugs (other than methotrexate).
  * Had received any intra-articular, intramuscular, or intravenous corticosteroids within 4 weeks prior to Baseline.
  * The subject had any previous use of cyclophosphamide, chlorambucil, or other alkylating agent.
* Was at high risk of an opportunistic infection because of a compromised immune system, in the investigator's opinion, with the exception of subjects receiving chronic steroid treatment.
* Had a history of or a current inflammatory condition with signs and symptoms that could have confounded the diagnosis of rheumatoid arthritis (eg, connective tissue disease, systemic lupus erythematosus, psoriasis, psoriatic arthritis, spondyloarthropathy).
* Had been diagnosed as having a secondary, non-inflammatory type of arthritis (eg, osteoarthritis or fibromyalgia) that, in the investigator's opinion, was symptomatic enough to interfere with the evaluation of the efficacy of the study drug on the subject's primary diagnosis of rheumatoid arthritis.
* Had a history of drug abuse or alcohol abuse within the past 2 years.
* The subject had a body mass index greater than 35 at Screening.
* Had a history of cancer, other than basal cell carcinoma, that had not been in remission for at least 5 years prior to the first dose of study drug.
* Had a known hypersensitivity to TAK-715 or its constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2004-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Composite ACR 20% improvement response rate from baseline with 3 of the following: pain assessment; disease activity; physical function; C-reactive protein and erythrocyte sedimentation rate. | Week 6

SECONDARY OUTCOMES:
Composite ACR 50% improvement response rate from baseline with 3 of the following: swollen-tender joint counts; pain assessment; disease activity; physical function; C-reactive protein and erythrocyte sedimentation rate. | Week 6.
Composite ACR 70% improvement response rate from baseline with 3 of the following: swollen-tender joint counts; pain assessment; disease activity; physical function; C-reactive protein and erythrocyte sedimentation rate. | Week 6.
Change from baseline in swollen and tender joint counts. | Week 6
Change from baseline in patient's assessment of pain. | Week 6
Change from baseline in patient's global assessment of disease activity. | Week 6
Change from baseline in physician's assessment of disease activity. | Week 6
Change from baseline in patient's self assessment of physical function using the Health Assessment Questionnaire. | Week 6
Change from baseline in C-reactive protein. | Week 6
Change from baseline in erythrocyte sedimentation rate. | Week 6
Time to American College of Rheumatology 20% improvement response. | Weeks 2, 4, and 6
Time to American College of Rheumatology 50% improvement response. | Weeks 2, 4, and 6
Time to American College of Rheumatology 70% improvement response. | Weeks 2, 4, and 6

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda